CLINICAL TRIAL: NCT06642376
Title: The Effect of Breathing Exercise Applied to Intensive Care Nurses on Fatigue and Perceived Stress: A Randomized Controlled Study
Brief Title: The Effect of Breathing Exercise Applied to Intensive Care Nurses on Fatigue and Perceived Stress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaraş İstiklal University (Other)
Responsible Party: Principal Investigator, Yasemin Sazak, Assistant Professor, Kahramanmaraş İstiklal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IstiklalU-YSazak-002
Record Dates: First submitted 2024-10-12; First posted 2024-10-15 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Breathing Exercises; Critical Care Nursing
Keywords: Stress; Nurse; Intensive care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing Exercise Application Group (Experimental): Nurses in the intervention group will be made to practice breathing exercises. The breathing exercise will first be explained to the nurses face-to-face and they will be made to do it. Then, face-to-face practice will be done three days a week, and on the other days, the audio recording of the breathing exercise will be sent by the researcher to the nurses via WhatsApp and they will be practiced daily. The breathing exercise will continue for 30 days.
  Interventions: Behavioral: Experimental: Breathing Exercise Application Group
- Control group (No Intervention): There will be no intervention for individuals in this group.

INTERVENTIONS:
Behavioral: Experimental: Breathing Exercise Application Group — The Effect of Breathing Exercise Applied to Intensive Care Nurses on Fatigue and Perceived Stress
  Arms: Breathing Exercise Application Group

SUMMARY:
The aim of this randomized controlled trial was to investigate the effect of breathing exercise on fatigue and stress in intensive care nurses.

Hypotheses of the study; H11: The level of perceived stress in nurses practicing breathing exercise is lower than the nurses in the control group.

H12: The level of fatigue is lower in nurses practicing breathing exercise compared to nurses in the control group.

Data will be collected in the intervention and control groups with a pre-test data collection form before the intervention. Patients in the intervention group will be given breathing exercises, while patients in the control group will not receive any intervention. In the second week, interim follow-up data will be collected with the data collection form. At the end of the study; data will be collected from the intervention and control groups with post-test data collection forms.

DETAILED DESCRIPTION:
In line with the randomization list, nurses will be assigned to the intervention and control groups in line with the inclusion criteria. The nurses will be informed about the study and their written and verbal consent will be obtained to participate in the study. Data will be collected from the nurses in the intervention and control groups with a pre-test data collection form. The nurses in the intervention group will be given breathing exercise practice, while the patients in the control group will not be subjected to any intervention. In the research; triple breathing technique (full yogic breathing) and 4-7-8 breathing technique will be used. In the intervention group, the nurses will first be told face-to-face about the breathing practice and have them do it. Then, face-to-face practice will be done three days a week, and on the other days, an audio recording of the breathing exercise will be sent by the researcher to the nurses via WhatsApp and they will be practiced daily. Breathing exercise will continue for 30 days in the intervention group. Follow-up data will be collected from the control and intervention group on the 15th day as an interim follow-up (with Piper fatigue scale and perceived stress scale). On the 30th day, the research will be finalized by collecting the post-test data. At the end of the study, the nurses in the control group will be shown and practiced breathing exercises.

ELIGIBILITY:
Inclusion Criteria:

* Working in intensive care for at least 6 months
* Volunteering to participate in the research
* Not practicing any complementary therapies during the study, such as breathing exercises, acupuncture, massage therapy, relaxation techniques and yoga, which may be effective on perceived stress and fatigue

Exclusion Criteria:

* Having a problem that prevents nasal breathing and prevents breathing exercises
* Being pregnant
* Experiencing physical and mental health problems that prevent communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Piper Fatigue Scale | 0 days
  The scale was developed by Piper et al. in 1987 to assess fatigue with the "integrated fatigue model". The Turkish validity and reliability study of the scale was conducted by Can et al. in 2004. The PMS consists of a total of 22 items, each rated on a 0-10 point Visual Analog Scale (VAS), and four sub-dimensions that assess the patient's subjective perception of fatigue.
Piper Fatigue Scale | 15 days
  The scale was developed by Piper et al. in 1987 to assess fatigue with the "integrated fatigue model". The Turkish validity and reliability study of the scale was conducted by Can et al. in 2004. The PMS consists of a total of 22 items, each rated on a 0-10 point Visual Analog Scale (VAS), and four sub-dimensions that assess the patient's subjective perception of fatigue.
Piper Fatigue Scale | 30 days
  The scale was developed by Piper et al. in 1987 to assess fatigue with the "integrated fatigue model". The Turkish validity and reliability study of the scale was conducted by Can et al. in 2004. The PMS consists of a total of 22 items, each rated on a 0-10 point Visual Analog Scale (VAS), and four sub-dimensions that assess the patient's subjective perception of fatigue.
Perceived Stress Scale | 0 days
  The Perceived Stress Scale was developed by Cohen, Kamarck and Mermelstein in 1983 and was designed to measure the extent to which people perceive the situations in their lives as stressful. The Turkish validity and reliability study of the scale was conducted by Mehmet Eskin et al. in 2013. It consists of 14 items and 2 sub-dimensions. In the 14-item perceived stress scale, scores range from 0 to 56. A high score in the questionnaire indicates a high perception of stress.
Perceived Stress Scale | 15 days
  The Perceived Stress Scale was developed by Cohen, Kamarck and Mermelstein in 1983 and was designed to measure the extent to which people perceive the situations in their lives as stressful. The Turkish validity and reliability study of the scale was conducted by Mehmet Eskin et al. in 2013. It consists of 14 items and 2 sub-dimensions. In the 14-item perceived stress scale, scores range from 0 to 56. A high score in the questionnaire indicates a high perception of stress.
Perceived Stress Scale | 30 days
  The Perceived Stress Scale was developed by Cohen, Kamarck and Mermelstein in 1983 and was designed to measure the extent to which people perceive the situations in their lives as stressful. The Turkish validity and reliability study of the scale was conducted by Mehmet Eskin et al. in 2013. It consists of 14 items and 2 sub-dimensions. In the 14-item perceived stress scale, scores range from 0 to 56. A high score in the questionnaire indicates a high perception of stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Istiklal Universty, Kahramanmaraş, Turkey (Türkiye)